CLINICAL TRIAL: NCT07245992
Title: A Dose-finding Phase I Study of F8IL10 Intra-articular Treatment in Rheumatoid Arthritis
Brief Title: A Study of F8IL10 Intra-articular Treatment in Rheumatoid Arthritis
Acronym: DekaJoint
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PH-F8IL10INTRA-03/24; 2024-517896-19-00 (EU CTIS Number)
Record Dates: First submitted 2025-08-19; First posted 2025-11-24 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: The dose escalation part of the study is designed with an accelerated phase, followed by a classical 3+3 dose escalation scheme.
  During the accelerated phase from 25 to 1000 μg F8IL10, cohorts contain one patient until the first instance of a treatment-related AE or DLT in the observation period from Day 1 - Day 28. With the occurrence of a treatment-related AE in the DLT observation period, two additional patients will be treated at the same dose level. If these two patients do not experience a treatment-related AE or a DLT, the accelerated phase of the study with initially one patient per dose level continues.
  With the second occurrence of a treatment-related AE (without DLT) within the observation period, the accelerated phase will be terminated, and the dose escalation part continues following the classical 3+3 design at the next higher dose level. With the first occurrence of a DLT in the DLT observation period, the dose escalation continues with the classical 3+3 design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): The study will take place in two stages:
  1. In the dose escalation part, participants will be enrolled in cohorts and will be treated with different dose levels of F8IL10 in order to identify a RD. In each cohort, 1 to 6 patients will be treated until the MAD is reached.
  2. Following successful identification of the RD, the study will proceed with a dose expansion part, during which 12 patients will be treated at RD (including those treated in the dose escalation part).
  Interventions: Drug: F8IL10

INTERVENTIONS:
Drug: F8IL10 — Intra-articular treatment

SUMMARY:
The aim of this study is to evaluate the safety of F8IL10 when administered by intra-articular injection and to determine the maximum tolerated dose (MTD) in order to establish the recommended dose (RD) in patients with Reumatoid Arthritis.

DETAILED DESCRIPTION:
This protocol describes an open-label, non-randomized, ascending dose, phase I study conducted in sequential cohorts of patients. The aim of the study is to assess the safety and tolerability of F8IL10 when administered via intra-articular (IA) route 3 times every 4 weeks in patients with RA.

Elegible patients of this trial are male or female, ≥ 18 and ≤ 80 years old, patients with Rheumatoid Arthritis (RA) who, despite treatment with stable doses (for at least 3 months) of DMARDs (conventional, biologic and/or targeted synthetic), present arthritis flare(s) suitable for IA injection in a knee, shoulder, ankle, wrist or elbow.

The study will take place in two stages:

1. The dose escalation part of the study is designed with an accelerated phase, followed by a classical 3+3 dose escalation scheme. Patients will be sequentially assigned to the following dose levels:

   * Cohort 1: 25 μg F8IL10
   * Cohort 2: 50 μg F8IL10
   * Cohort 3: 100 μg F8IL10
   * Cohort 4: 400 μg F8IL10
   * Cohort 5: 700 μg F8IL10
   * Cohort 6: 1000 μg F8IL10
2. Following successful identification of the RD, the study will proceed with a dose expansion part, during which 12 patients will be treated at RD (including those treated in the dose escalation part).

Patients will receive intra-articular administations of F8IL10 every 4 weeks for up to 3 administrations.

Following completion of the treatment, patients will continue with Follow-up for up to 6 months (Week 37) to monitor the duration of treatment response as well as their health status, the possible onset of post-treatment AEs and the modifications to the treatment that may be required to manage disease symptoms, if any.

The primary objective is to evaluate the safety of F8IL10 when administered by IA injection and to determine the maximum tolerated dose (MTD) in order to establish the recommended dose (RD).

Secondary objectives are to assess early signs of efficacy and to determine the pharmacokinetic profile and immunogenicity of intra-articular F8IL10.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 and ≤80 years.
2. Diagnosis of RA according to ACR/EULAR classification criteria (2010) with a disease duration exceeding 6 months.
3. Presence of arthritis flare(s) suitable for IA injection in a knee, ankle, shoulder, wrist or elbow, despite treatment with stable doses (for at least 3 months) of DMARDs (conventional, biologic, and targeted synthetic) background therapy.
4. No or stable regimens of NSAIDs and/or oral corticosteroid (≤ 10 mg/day; prednisone equivalent) for a period ≥2 weeks prior to screening.
5. All acute toxic effects of any prior therapy must have resolved or returned to classification "mild" (grade 1) according to CTCAE v.5.0.
6. Sufficient hematologic, liver and renal function defined as follows:

   * Absolute neutrophil count (ANC) ≥1.5 x 109/L, platelets ≥100 x109/L, haemoglobin (Hb) ≥10.0 g/dL.
   * Alkaline Phosphatase (AP), Alanine Aminotransferase (ALT) and or Aspartate Aminotransferase (AST) ≤3 x Upper Limit of Normal Range (ULN), and total bilirubin ≤2.0 mg/dl (34.2 μmol/L).
   * Creatinine ≤1.5 ULN or 24 h creatinine clearance ≥50 mL/min.
7. Documented negative TB test (e.g. Quantiferon or equivalent).
8. Documented negative test for HIV-HBV-HCV. For HBV serology, the determination of HBsAg and anti-HBcAg Ab is required. In patients with serology documenting previous exposure to HBV (i.e., anti-HBs Ab with no history of vaccination and/or anti-HBc Ab), negative serum HBV-DNA is required. For HCV, HCV-RNA or HCV antibody test is required. Subjects with a positive test for HCV antibody but no detection of HCV-RNA indicating no ongoing infection are eligible.
9. Sexually active male or female patients of childbearing potential are eligible providing that:

   * Women of childbearing potential (WOCBP) have a negative pregnancy test performed within 4 weeks prior to treatment start.
   * WOCBP agree to use, from the screening to 6 months following the last study drug administration, effective method of birth control as applicable per local law that both results in a Pearl index <1 and considered highly effective as defined by the "Recommendations for contraception and pregnancy testing in clinical trials" issued by the "Clinical Trial Facilitation Group" (e.g. combined estrogen and progestogen containing hormonal contraception, progestogen-only hormonal contraception, intrauterine device, intrauterine hormone-releasing system, vasectomized partner, total sexual abstinence or bilateral tubal occlusion).
   * Males agree to use two acceptable methods of contraception (e.g. condom with spermicidal gel) from the screening to 6 months following the last study drug administration. Females of childbearing potential that are partners of male study participants must observe the same birth control indications that apply to female participants.
10. Signed and dated Ethics Committee-approved informed consent form indicating that the patient, or patient's legally acceptable representative, has been informed of all pertinent aspects of the study.
11. Willingness and ability to comply with the scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Presence of additional RA flares or RA-related symptoms that, in the investigator's judgment, are likely to require local treatment during the study (defined as intra-articular or peri-articular injections/procedures intended to treat RA; e.g., joint, tendon-sheath, or bursal corticosteroid injections; hyaluronic acid; biologic/PRP injections; or radio synovectomy)._
2. Presence of active infections or another severe concurrent disease, which, in the opinion of the investigator, would place the patient at undue risk or would interfere with the study objectives or conduct.
3. Pregnancy, lactation or unwillingness to use adequate contraceptive methods.
4. Diagnosis of any other inflammatory arthritis or active autoimmune diseases other than RA.
5. Any therapy for RA apart from the allowed background therapy (i.e., stable doses of DMARDs, corticosteroids, and/or NSAIDs) within 4 weeks prior to the first IMP dosing.
6. Received intra-articular administration of corticosteroids/DMARDs within 4 weeks or 5 half-lives prior to the first IMP dosing, whichever is longer.
7. History or currently active primary or secondary immunodeficiency.
8. Concurrent malignancy or history of malignancy (except in situ melanoma and low-risk non melanoma skin cancer) from which the patient has been disease-free for less than 2 years.
9. History within the last year of acute or subacute coronary syndromes including myocardial infarction, unstable or severe stable angina pectoris.
10. Treatment with warfarin or other coumarin derivatives.
11. Clinically significant cardiac arrhythmias or requiring permanent medication.
12. Abnormalities in baseline ECG analysis that are considered as clinically significant by the investigator; subjects with current or a history of QT/QTc prolongation.
13. Uncontrolled hypertension, despite optimal treatment.
14. Known arterial aneurism at high risk of rupture.
15. Ischemic peripheral vascular disease (Grade IIb-IV according to Leriche Fontaine classification).
16. Severe diabetic retinopathy.
17. Major trauma including surgery within 4 weeks prior to administration of study treatment.
18. Known history of allergy/hypersensitivity or other intolerance to any component of F8IL10 (including excipients) or to other drugs based on human proteins/peptides/antibodies.
19. Treatment with any investigational agent within 4 weeks or 5 half-lives prior to the first dose of study drug, whichever is longer.
20. Immunization with a live/attenuated vaccine within 4 weeks prior to baseline or plan to receive vaccines during the study.
21. Non-RA related chronic pain disorders.
22. Patients requiring stable doses of corticosteroids >10 mg/day (prednisone equivalent). Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions is not considered an exclusion criterion.
23. History of alcohol, drug or chemical substance abuse within the 6 months prior to screening.
24. Any condition that in the opinion of the investigator could hamper compliance with the study protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
DLT | From Day 1 to Day 28 of the treatment
  Occurrence of dose limiting toxicity (DLT)
MAD, MTD and RD | From Day 1 to Day 28 of the treatment
  Definition of maximum administered dose (MAD), maximum tolerated dose (MTD) and recommended dose (RD)
AEs, SAEs and DILI | Through study completation (up to 37 weeks)
  Adverse events (AEs), serious adverse events (SAEs) and Drug-Induced Liver Injury (DILI), based on Common Terminology Criteria for Adverse Events v. 5.0 (CTCAE).
Incidence of injection site reactions | Through study completation (up to 37 weeks)
  Incidence of injection site reactions and general reactions associated with intraarticular administration
Standard laboratory parameters | Through study completion (up to 37 weeks)
  Standard laboratory (haematology, biochemistry, liver and urine analysis) parameters.

SECONDARY OUTCOMES:
CCI: Composite change index | Every 4 weeks, up to week 37
  The CCI is a semiquantitative scoring system designed to assess target joint synovitis by integrating multiple clinical variables. It incorporates changes in joint pain measured by the Visual Analogue Scale (jVAS), clinical evaluation of joint swelling and tenderness, the patient's assessment of functional disability, and both patient and investigator global assessments of treatment efficacy. The resulting score ranges from 0 (no improvement) to 10 (maximal therapeutic effect).
SF-36 | Every 4 weeks, up to week 37
  Changes in Short Form Health Survey 36. The SF-36 is a validated, patient-reported measure of overall health status, comprising multi-item scales measuring each of the following 8 health concepts: (1) physical functioning, (2) role limitations due to physical health, (3) bodily pain, (4) social functioning, (5) emotional well-being, (6) role limitations due to emotional problems, (7) vitality (energy/fatigue), and (8) general health perceptions. Each healt concept is scored separately, with scores ranging from 0 (worst possible health status) to 100 (best possible health status).
Joint inflammation | Every 4 weeks, up to week 37
  Changes in target joint inflammation (synovitis) assessed by gray-scale ultrasound (GSUS) and power doppler ultrasound (PDUS). Ultrasound assessment of the treated joint will be performed using gray-scale (to evaluate hypoechoic synovial hypertrophy) and power Doppler (to assess synovial vascularity). Semiquantitative scoring will be applied to each modality separately, as well as in a combined score, ranging from grade 0 (normal) to grade 3 (severe synovitis).
SDAI | Every 4 weeks, up to week 37
  Changes in Simple Disease Activity Index. The SDAI is a validated tool for assessing rheumatoid arthritis disease activity. It sums the tender and swollen joint counts, patient and physician global assessments of disease activity, and C-reactive protein levels in serum. Scores indicate disease activity: ≤3.3 (remission), >3.3-11 (low), >11-26 (moderate), and >26 (high).
Pharmacokinetic profile | Every 2 weeks, up to week 7
  Pharmacokinetic profile of intra-articular F8IL10.
HAFA | Every 4 weeks, up to week 17
  Formation of human anti-fusion protein antibodies (HAFA) against F8IL10.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Arcispedale Santa Maria Nuova, Reggio Emilia, Reggio Emilia
  - Azienda Ospedaliera Universitaria Integrata Verona c/o Policlinico GB Rossi (Borgo Roma), Dep. Reumatologia, Verona, VR

IPD SHARING:
Plan to Share IPD: No